CLINICAL TRIAL: NCT01168440
Title: A Single-arm, Phase II Study of Sunitinib in Patients With Von Hippel-Lindau (VHL) Disease
Brief Title: Study of Sunitinib in Patients With Von Hippel-Lindau (VHL) Disease
Acronym: VHLSUT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Pr Stephane OUDARD, MD, PhD, ARTIC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHLSUT09
Record Dates: First submitted 2010-03-18; First posted 2010-07-23 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Von Hippel-Lindau Disease
Keywords: von Hippel-Lindau; VHL; sunitinib
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sunitinib — Sunitinib, 50 mg PO daily, 6 weeks courses with schedule 4/2 (4 weeks of treatment followed by 2 weeks of rest).

SUMMARY:
VHL patients may benefit from sunitinib. This study will investigate the following objectives :

PRIMARY OBJECTIVE

* To determine the objective response rate according to RECIST criteria, in VHL patients with advanced tumors or tumors untreatable by other means, and treated with sunitinib.

SECONDARY OBJECTIVES

* To evaluate the safety and tolerability of sunitinib in VHL patients according to the NCI-CTC criteria Version 3.0.
* To determine the following time-to-event endpoints: overall survival, time to disease progression, progression free survival, time to response and duration of response.
* To evaluate quality of life in VHL patients receiving sunitinib.

DETAILED DESCRIPTION:
Treatment with sunitinib, 50 mg PO daily, 6 weeks courses with schedule 4/2 (4 weeks of treatment followed by 2 weeks of rest).

Treatment until disease progression or unacceptable toxicity.

Dose reduction depending on type and severity of toxicity. At the end of treatment period (after 8 courses), responding and well tolerating patients will be allowed to receive sunitinib upon investigator's opinion.

Follow-up for up to 24 months from inclusion.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients must have genetically or clinically confirmed VHL disease and have symptoms from VHL that are no longer controllable by conventional approaches.
2. Patients must have at least one of the following lesions :

   * Eye : retinal hemangioblastoma that can no longer be treated by laser therapy or cryotherapy and resulting in progressive loss of vision;
   * CNS : cerebellar, bulbar, spinal, or cerebellopontine angle haemangioblastoma or endolymphatic sac tumor causing neurological symptoms that are not amenable to further surgery, or have recurred after a first surgery;
   * Kidney: multiple or bilateral tumors not accessible to conservative surgery, or tumors having recurred after surgery and/or radiofrequency ablation or advanced/metastatic RCC;
   * Pancreas: inextirpable or advanced neuroendocrine tumors.
3. Patients previously treated for VHL with surgery, chemotherapy or radiotherapy are considered eligible for this study under the condition that these treatments were completed more than 4 weeks prior starting the study treatment. Previously radiated lesions will be considered as target lesions only if they demonstrate unequivocal evidence of growth upon imagery.
4. Male or female, at least 18 year-old.
5. Performance status ECOG 0-2
6. Life expectancy = 3 months
7. Biological/clinical values within the following limits:

   * Total serum bilirubin = 1.5 x ULN (patients with Gilbert's disease are not eligible)
   * Serum transaminases and alkaline phosphatases = 2.5 x ULN, or in case of underlying malignancy (hepatic metastasis) = 5x ULN
   * Serum creatinine = 1.5 x ULN, creatinine clearance = 80 ml/min
   * Absolute neutrophil count = 1500/mm3
   * Platelets = 100,000/mm3
   * Hemoglobin = 9.0 g/dL
   * QTc interval = 450 msec
   * Left ventricular ejection fraction (LVEF) = lower limit of institutional normal as assessed by multigated acquisition (MUGA) scan or echocardiogram
8. Eligibility of patients receiving any medications or substances which may alter the activity or pharmacokinetics of sunitinib (CYP3A4 inhibitors or inducers among which ketoconazole, theophylline, phenobarbital, coumadin/warfarin) will be decided after review by the principal investigator of possibility to interrupt or switch to other medications. Otherwise, patient is not eligible. Anticoagulants drugs (among which coumadin/warfarin) may be, either switched to low-molecular-weight heparin, or be subject to individual dose adaptation in order to maintain INR in the target range with regard to patient's history, all along his participation in the study.
9. Signed and dated informed consent document stating that the patient, or legally representative, has been informed of all the aspects of the trial prior to enrollment
10. Willingness and ability to comply with all protocol assessments, schedule of visits, and procedures that are or could be requested as part of this study.
11. Affiliated to French social security system

EXCLUSION CRITERIA

1. Chemotherapy, radiotherapy, radiofrequency or surgery within 4 weeks prior to entering the study or not complete recovering from adverse events due to drugs administered more than 4 weeks earlier.
2. Patients receiving any other investigational agent or having participated in a clinical trial in the last 30 days.
3. History of allergic reaction attributed to compounds of similar chemical or biological composition to sunitinib.
4. Previous treatment with sunitinib
5. NCI-CTCAE grade = 3 hemorrhage within 4 weeks prior to study entry.
6. History of known or suspected brain metastases, spinal cord compression, carcinomatous meningitis, evidence of leptomeningeal disease (excepted leptomeningeal hemangioblastoma, according to the neurologist) on screening CT scan or MRI.
7. Any of the following within the 6 months prior to study drug administration: symptomatic congestive heart failure, myocardial infarction or coronary artery bypass, pulmonary embolism, ongoing severe or unstable angina pectoris, NCI-CTCAE grade = 2 cardiac dysrhythmia, cerebrovascular accident or transient ischemic attack.
8. Hypertension >140/90 mmHg that cannot be controlled despite optimal antihypertensive therapy.
9. Pre-existing thyroid abnormality with thyroid function that cannot be maintained in the normal range despite medication.
10. Other severe acute or chronic medical condition including (but not limited to), ongoing infection, unstable or uncompensated respiratory, cardiac, hepatic or renal disease, psychiatric condition, laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which would make the patient inappropriate for entry into the trial.
11. Any medical condition (gastric or small intestine pathology, malabsorption syndrome) that might interfere with oral medication absorption.
12. Known HIV-positive patients treated with antiretroviral therapy (potential pharmacokinetic interactions with sunitinib).
13. Pregnancy or breastfeeding. Patients must agree to use effective contraception during the study, including oral contraceptives, intrauterine devices, or being unable to procreate.
14. Any other malignancy within the last 3 years excepted basal cell carcinoma, in situ cervical carcinoma, squamous cell skin cancer, pT1/a bladder cancer with no evidence of recurrence during the last 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Objective response rate (RECIST criteria) | Every 6 weeks
  Course: 4 weeks sunitinib / 2weeks rest. Response assessment: after 4 weeks and 8 weeks of sunitinib (1 extra assessment by contrast-enhanced US after 2 weeks for kidney tumors). Then every 6 weeks for eye and every 12 weeks for all other tumors.

SECONDARY OUTCOMES:
Safety and tolerability (NCI-CTC criteria Version 3.0). | Every 6 weeks
Time-to-event endpoints: overall survival, time to disease progression, progression free survival, time to response and duration of response. | Every 6 weeks
Quality of life in VHL patients receiving sunitinib. | Every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephane RICHARD, MD, PhD, Principal Investigator — Hôpital Kremlin-Bicêtre (France); Reza T ELAIDI, PhD, Study Director — ARTIC (Hopital Européen Georges Pompidou, FRANCE)
Locations (3):
- France (3):
  - Hospital Saint André - Service de cancérologie, Bordeaux
  - Hopital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Européen Georges Pompidou - Service d'Oncologie Médicale, Paris